CLINICAL TRIAL: NCT01207960
Title: A Randomized Wait-list Control Study of the Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) in Patients With Dental Phobia
Brief Title: Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) in Dental Phobia
Acronym: EMDR-DP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, doerings, Univ.-Prof. Dr., University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-137-f-S
Record Dates: First submitted 2010-06-29; First posted 2010-09-23 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Dental Phobia
Keywords: dental phobia; psychotherapy; eye movement desensitization and reprocessing - EMDR; efficacy; wait-list control
MeSH Terms: interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMDR (Active Comparator): Eye Movement Desensitization and Reprocessing
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)
- WLC (No Intervention): Wait-list control group. EMDR treatment takes place after 4 weeks of no treatment which represents the wait-list comparison interval.

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) — The intervention consists of three 90-minute sessions of individual psychotherapy. Sessions take place weekly according to a treatment manual.
  Arms: EMDR

SUMMARY:
The purpose of this study is to find out whether Eye Movement Desensitization and Reprocessing (EMDR) is effective in the treatment of patients with dental phobia.

DETAILED DESCRIPTION:
Dental phobia represents a clinical condition that affects 5-15% of the community and is characterized by severe anxiety of dental treatment which leads to avoidance of treatment and, as a consequence, severe dental as well as psychosocial problems.

Eye Movement Desensitization and Reprocessing (EMDR) has been developed for the treatment of patients with post traumatic stress disorder (PTSD). Its efficacy in PTSD patients has often been demonstrated in randomized controlled trials.

Recently it has been demonstrated that dental phobia is often induced by traumatic events during dental treatment and goes along with symptoms of PTSD in numerous patients.

A pilot study (de Jongh et al. 2002) gave hints on the efficacy of EMDR in four dental phobia patients with a history of traumatization during dental treatment.

This randomized wait-list control study aims to evaluate the efficacy of EMDR in a larger sample of dental phobia patients.

ELIGIBILITY:
Inclusion Criteria:

* dental phobia according to the World Health Organization´s International Classification of Diseases, ICD-10 (F40.2)

Exclusion Criteria:

* schizophrenic disorder
* severe depression
* severe dissociative disorder
* organic brain disease
* anorexia nervosa (body mass index, BMI < 17)
* suicidality
* severe cardio-vascular disease
* ophthalmic disease
* pregnancy and lactation
* psychopharmacological treatment
* substance abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Dental anxiety | 4 weeks
  Dental anxiety is assessed by the Dental Anxiety Scale (DAS) and the Dental Fear Survey (DFS).
Dental anxiety | 3 months
  Dental anxiety is assessed by the Dental Anxiety Scale (DAS) and the Dental Fear Survey (DFS).
Dental anxiety | 12 months
  Dental anxiety is assessed by the Dental Anxiety Scale (DAS) and the Dental Fear Survey (DFS).

SECONDARY OUTCOMES:
General psychopathology | 4 weeks, 3 months, 12 months
  General psychopathology is assessed by the Brief Symptom Scale (BSI).
Anxiety and depression | 4 weeks, 3 months, 12 months
  Anxiety and depression are assessed by the Hospital Anxiety and Depression Scale (HADS).
Behavioral test | 4 weeks
  Dentral anxiety is assessed during a dental visit before and after treatment/wait-list control condition by means of a standardized behavior obeservation and interview.
Dental treatment | 3 months, 12 months
  Does the patient tolerate dental treatment within 3 and 12 months after Eye Movement Desensitization and Reprocessing (EMDR)?

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Doering, MD, Principal Investigator — University of Muenster, Germany
Locations (1):
- Psychosomatics in Dentistry, Dept. of Prosthodontics & Material Science, University Hospital Muenster, Münster, Germany

REFERENCES:
- [Background] De Jongh A, van den Oord HJ, ten Broeke E. Efficacy of eye movement desensitization and reprocessing in the treatment of specific phobias: Four single-case studies on dental phobia. J Clin Psychol. 2002 Dec;58(12):1489-503. doi: 10.1002/jclp.10100. PMID 12455017
- [Background] de Jongh A, Fransen J, Oosterink-Wubbe F, Aartman I. Psychological trauma exposure and trauma symptoms among individuals with high and low levels of dental anxiety. Eur J Oral Sci. 2006 Aug;114(4):286-92. doi: 10.1111/j.1600-0722.2006.00384.x. PMID 16911099